CLINICAL TRIAL: NCT02075996
Title: Non-interventional Study of Pomalidomide (Imnovid®) in Combination With Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Non-interventional Study With Pomalidomide (Imnovid®)
Acronym: Poseidon
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-10280
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Multiple Myeloma
Keywords: pomalidomide, Imnovid, dexamethasone, Poseidon, multiple myeloma, daily routine, secondary malignancies, Germany, non-interventional study, safety,
MeSH Terms: conditions — Multiple Myeloma; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pomalidomide following lenalidomide: 75 patients with pomalidomide directly following lenalidomide treatment
- Pomalidomide following other therapy: 75 patients with pomalidomide following any other prior therapy. This includes lenalidomide in earlier lines than the most recent line.

SUMMARY:
The purpose of this non-interventional study is to collect data on the efficiency and safety of pomalidomide in combination with dexamethasone in the routine application

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory multiple myeloma Patients must have received at least two prior lines of treatment (induction therapy followed by stem cell transplantation ± maintenance therapy is considered one prior therapy) and must have progressed under the most recent therapy regimen
* Adult male and female patients (at least 18 years with no upper age limit)
* Written informed consent to data collection and pseudonymized data transfer
* The conditions of the Pregnancy Prevention Programme must be fulfilled for all patients unless there is reliable evidence that the patient does not have childbearing potential (see summary of product characteristics Imnovid®)
* Other criteria according to summary of product characteristics Imnovid®

Exclusion Criteria:

* Missing patient's informed consent
* Pregnant or breast-feeding women
* Male patients, not capable of complying the required preventive measures (see summary of product characteristics Imnovid®)
* Other criteria according to summary of product characteristics Imnovid®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with relapsing or refractory multiple myeloma previously treated with at least two prior lines of therapy, including bortezomib and lenalidomide who have progressed under their last therapy regimen
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2014-02-11 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 6 years

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 6 years
Time to Treatment Discontinuation (TTD) | 6 years
Time to next treatment (TNT) | 6 years
adverse reaction profile | 3 years
secondary malignancies | 6 years
  long term safety is focused on secondary malignancies
overall Survival (OS) | 6 years
relative dose intensity of pomalidomide and dexamethasone | 3 years
assess changes in myeloma-related quality of life | 3 years
explore additional supportive therapies | 3 years
  To explore additional supportive therapies used on this patient population (e.g. G-CSF, antibiotics, DVT prophylaxis)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Dechow, PhD, Principal Investigator — practice based oncology office Ravensburg
Locations (1):
- iOMEDICO AG, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Dechow T, Aldaoud A, Behlendorf T, Knauf W, Eschenburg H, Groschek M, Hansen R, Soling U, Grebhardt S, Siebenbach HU, Vannier C, Potthoff K. Pomalidomide plus dexamethasone for patients with relapsed or refractory multiple myeloma: Final results of the non-interventional study POSEIDON and comparison with the pivotal phase 3 clinical trials. Eur J Haematol. 2022 Feb;108(2):133-144. doi: 10.1111/ejh.13719. Epub 2021 Nov 15. PMID 34714555